CLINICAL TRIAL: NCT06673147
Title: Effects of Nordic Walking on Prenatal Health: A Focus on Gait Kinematics, Musculoskeletal Pain, and Quality of Life. A Randomized Controlled Trial.
Brief Title: Effects of Nordic Walking on Prenatal Health
Acronym: Nordic Walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Wafaa Mahmoud Amin, Lecturer, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RHPT/024/016; RHPT/024/016 (Other: Prince Sattam bin Abdulaziz University)
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2024-11

CONDITIONS: Prenatal Care; Walking
Keywords: Prenatal health Nordic walking; pregnancy; musculoskeletal pain; gait parameters; quality of life
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Out of 50 pregnant women who will be screened for their eligibility criteria, The participants will be randomized to either intervention group (Nordic Walking) or control group (standard prenatal care).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): It will be receiving Nordic walking training
  Interventions: Other: Prenatal Nordic Walking
- Control Group (No Intervention): This group will receive a standard prenatal care, which included routine obstetric check-ups and general advice on physical activity

INTERVENTIONS:
Other: Prenatal Nordic Walking — Traditional Nordic walking poles will be modified according to International Nordic Walking Federation guidelines, which meant that the elbows were bent at a 90°angle when holding the poles in a vertical position. Nordic Walking will be conducted in two phases consisting of a 4-week learning phase followed by an 8-week main phase of intervention.
  Arms: Intervention group

SUMMARY:
This randomized controlled trial (RCT) aimed to evaluate the effects of Nordic walking (NW) on gait kinematics, musculoskeletal pain, and quality of life in pregnant women.

DETAILED DESCRIPTION:
Healthy pregnant women (N=50), aged 20-40 years and between 13 and 28 weeks of gestation, experiencing mild to moderate musculoskeletal pain, will be recruited. Participants will be randomized into either an intervention group (NW training) or a control group receiving standard prenatal care. The intervention group will undergo a 4-week learning phase followed by an 8-week NW program (3 sessions per week, 45 minutes per session), led by a certified instructor. Outcome measures will be assessed at baseline, after 4 weeks, and post-intervention (8 weeks), including spatiotemporal gait parameters (will be assessed using the GAITRite system), musculoskeletal pain (will be measured via Visual Analog Scale, VAS), and quality of life (will be measured using the SF-36 Health Survey).

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 20 to 40 between 13 and 28 weeks into singleton pregnancy.
* Participants must be experiencing mild to moderate musculoskeletal discomfort, such as lower back or pelvic pain,
* Participants have no prior musculoskeletal or neurological diseases.
* They must have no contraindications to exercising throughout pregnancy, as established by obstetrician clearance, and be able to engage in moderate physical activity under medical recommendations

Exclusion Criteria:

* History of diseases affecting bony structures or lumbar intervertebral discs.
* Pain caused by non-musculoskeletal factors (such as urinary tract infections or obstetric complications).
* Multiple pregnancies, pre-existing mobility conditions, and high-risk pregnancies or complications that restrict physical activity.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-06-29 (Actual)

PRIMARY OUTCOMES:
Spatial gait parameters | 20 minutes
  A GAITRite system will be used to assess the spatial parameters of gait
Temporal parameters of gait | 20 minutes
  A GAITRite system will be used to assess the temporal parameters of gait

SECONDARY OUTCOMES:
Visual Analog Score for musculoskeletal pain | 5 minutes
  The Visual Analog Score is depicted as a 10 cm horizontal line divided into 1 cm sections, each representing 1 point, resulting in a score ranging from 0 to 10 points. Higher scores mean worse outcome.
Quality of life | 10 minutes
  The SF-36 Health Survey will be used to determine the results.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia L Radwan, PHD, Study Director — Prince Sattam Bin Abdulaziz University
Locations (1):
- Department of Health and Rehabilitation Sciences, Prince Sattam bin Abdulaziz University., Riyadh, Alkharj, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No